CLINICAL TRIAL: NCT03675971
Title: COPE: Cannabinoids to Obviate Pain Experiment After Knee Replacement
Acronym: COPE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCT19-366965
Record Dates: First submitted 2018-08-28; First posted 2018-09-18 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Pain Management; Analgesics, Opioid; Cannabis
MeSH Terms: conditions — Agnosia; Marijuana Abuse | interventions — Cannabinol; Medical Marijuana

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Cannabis (Experimental): Drug: Cannabidiol
  Interventions: Drug: Cannabinol
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Cannabinol — Postoperative pain treatment
  Other Names: medical cannabis
  Arms: Medical Cannabis
Drug: Placebo oral capsule — Placebo comparator
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Total knee replacement is a major and painful orthopaedic (joint and bone) surgery where the knee joint is replaced with an artificial joint. It is an effective and successful procedure to treat severe knee arthritis and reduce pain, but many patients report intense pain after the surgery.

Postoperative pain control is predominated by opioids (morphine-based drugs). While opioids are effective to manage the pain, they can have acute and chronic complications, including confusion, nausea, vomiting, constipation and high risk of addiction.

Medical cannabis is an effective and safe alternative for pain treatment. Recent studies showed that patients have reported a reduction in opioid usage when taking cannabis as a substitute for pain relief.

This study aims to investigate whether adding medical cannabis (cannabidiol - CBD) treatment will decrease the amount of opiates needed in the first 2 weeks after knee replacement compared to a group given placebo.

DETAILED DESCRIPTION:
COPE (Cannabinoids to Obviate Pain Experiment after knee replacement) will be a single-centre, prospective, randomized, placebo-controlled, superiority trial, with two parallel groups designed to investigate the effect of cannabis as postoperative pain treatment compared to placebo on total opioid consumption after total knee replacement.

Eligible patients are: men and non-pregnant women aged ≥18 years scheduled to undergo primary total knee replacement. and with no opioid usage within the last 3 months or history of narcotic abuse.

Patients will be recruited at the department of orthopaedic surgery at St Michael's Hospital (Toronto - Canada), and informed consent will be obtained from those eligible. Central computer-generated randomization will be used to randomly assign participants to cannabis or placebo groups (1:1 ratio). Only the study pharmacist will know allocated treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Men and women
* Patients with radiographic confirmation and clinical correlation for severe osteoarthritis diagnosis with an indication for total knee replacement
* Patients undergoing primary unilateral total knee replacement
* Patient is able to provide informed consent to participation in the study

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Current opioid use
* Cognitive impairment or mental illness (e.g., dementia, Alzheimer disease and psychoses), which will prevent patients from reliably providing primary outcome data
* Unable to swallow an oral tablet (medication)
* History of opiate, narcotic and alcohol abuse
* Revision total knee replacement surgery
* High risk of falls as determined by the treating physician
* Patients refusing participation
* Pre-existing/ regular cannabis use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 2 weeks after total knee replacement
  Assess cumulative opioid consumption (morphine equivalent dose) by means of drug reconciliation (medication diaries and pill counts) i.e. patients will self report how many opioid pills they took each day, by means of the medication diaries and at 4 weeks follow up will bring the pills back to clinic appointment.

SECONDARY OUTCOMES:
Visual Analog Pain Scale | Pain scale will be assessed at 24 hours, 2, 6 and 12 weeks after knee replacement
  Assess pain from a visual scale that ranges from 0 to 10. Straight line with the endpoints defining extreme limits such as 'no pain at all' (zero) and 'pain as bad as it could be' (ten)
Oxford knee score | Questionnaire will be completed by patients at 6 weeks after knee replacement
  A short questionnaire consists of 12 questions ranging from 0 to 48 points, designed to assess function and pain after knee replacement surgery. Higher values represent a better outcome. Scores between 40-48 indicate satisfactory joint function
Health status and quality of life | Questionnaire will be completed by patients at 6 weeks after knee replacement
  EQ-5D is a questionnaire where patients self-rate their level of severity of health status and health-related quality of life. Consists of 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and each one of them has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems) where patients will indicate how they feel regarding their health status and quality of life.
Quality of recovery - 15 (QoR-15) | Questionnaire will be completed by patients at 12 weeks after knee replacement
  Quality of recovery scores are patient-reported outcome measures evaluating recovery after surgery regarding the last 24h. It is a short-form score with 15 questions that assess the 5 dimensions (pain, physical comfort, physical independence, physiological support and emotional state) and has 2 parts (A and B). Part A scores from 0 [poor] to 10 [excellent] - as higher is the score as better is the recovery. Part B scores from 10 [excellent] to 0 [poor] - as higher is the score as better is the recovery.
Self-reported opioid use and urinalysis | The test will be completed at 12 weeks after knee replacement
  Patients will self report whether they are still using opioids (yes or no) and they will undergo a urinalysis (urine test). Patients will pee in a designed cup and a trained assessed will test the urine (with chemical strip) to detect the presence of one or more opioids in urine.
Narcotic monitoring prescription | Will be assessed at 12 months after knee replacement
  Using data from the Narcotics Monitoring System from ICES (Institute for Clinical Evaluative Sciences) which already captures all opioid prescriptions dispensed in retail pharmacies across Ontario, the investigators will assess if participants have had any filled prescription after knee replacement and record the number of prescriptions filled.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Atrey, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Institute for Health Information. Hip and Knee Replacements in Canada, 2016-2017: Canadian Joint Replacement Registry Annual Report. Ottawa, ON: CIHI; 2018
- [Background] Terkawi AS, Mavridis D, Sessler DI, Nunemaker MS, Doais KS, Terkawi RS, Terkawi YS, Petropoulou M, Nemergut EC. Pain Management Modalities after Total Knee Arthroplasty: A Network Meta-analysis of 170 Randomized Controlled Trials. Anesthesiology. 2017 May;126(5):923-937. doi: 10.1097/ALN.0000000000001607. PMID 28288050
- [Background] Canata GL, Casale V, Chiey A. Pain management in total knee arthroplasty: efficacy of a multimodal opiate-free protocol. Joints. 2017 Feb 7;4(4):222-227. doi: 10.11138/jts/2016.4.4.222. eCollection 2016 Oct-Dec. PMID 28217658
- [Background] Mohamadi A, Chan JJ, Lian J, Wright CL, Marin AM, Rodriguez EK, von Keudell A, Nazarian A. Risk Factors and Pooled Rate of Prolonged Opioid Use Following Trauma or Surgery: A Systematic Review and Meta-(Regression) Analysis. J Bone Joint Surg Am. 2018 Aug 1;100(15):1332-1340. doi: 10.2106/JBJS.17.01239. PMID 30063596
- [Background] Hadlandsmyth K, Vander Weg MW, McCoy KD, Mosher HJ, Vaughan-Sarrazin MS, Lund BC. Risk for Prolonged Opioid Use Following Total Knee Arthroplasty in Veterans. J Arthroplasty. 2018 Jan;33(1):119-123. doi: 10.1016/j.arth.2017.08.022. Epub 2017 Aug 24. PMID 28927564
- [Background] Morris BJ, Mir HR. The opioid epidemic: impact on orthopaedic surgery. J Am Acad Orthop Surg. 2015 May;23(5):267-71. doi: 10.5435/JAAOS-D-14-00163. PMID 25911660
- [Background] Goesling J, Moser SE, Zaidi B, Hassett AL, Hilliard P, Hallstrom B, Clauw DJ, Brummett CM. Trends and predictors of opioid use after total knee and total hip arthroplasty. Pain. 2016 Jun;157(6):1259-1265. doi: 10.1097/j.pain.0000000000000516. PMID 26871536
- [Background] Franklin PD, Karbassi JA, Li W, Yang W, Ayers DC. Reduction in narcotic use after primary total knee arthroplasty and association with patient pain relief and satisfaction. J Arthroplasty. 2010 Sep;25(6 Suppl):12-6. doi: 10.1016/j.arth.2010.05.003. Epub 2010 Jun 26. PMID 20580191
- [Background] Soffin EM, Waldman SA, Stack RJ, Liguori GA. An Evidence-Based Approach to the Prescription Opioid Epidemic in Orthopedic Surgery. Anesth Analg. 2017 Nov;125(5):1704-1713. doi: 10.1213/ANE.0000000000002433. PMID 29049115
- [Background] Cozowicz C, Olson A, Poeran J, Morwald EE, Zubizarreta N, Girardi FP, Hughes AP, Mazumdar M, Memtsoudis SG. Opioid prescription levels and postoperative outcomes in orthopedic surgery. Pain. 2017 Dec;158(12):2422-2430. doi: 10.1097/j.pain.0000000000001047. PMID 28891865
- [Background] Lynch ME, Campbell F. Cannabinoids for treatment of chronic non-cancer pain; a systematic review of randomized trials. Br J Clin Pharmacol. 2011 Nov;72(5):735-44. doi: 10.1111/j.1365-2125.2011.03970.x. PMID 21426373
- [Background] Schrot RJ, Hubbard JR. Cannabinoids: Medical implications. Ann Med. 2016;48(3):128-41. doi: 10.3109/07853890.2016.1145794. Epub 2016 Feb 25. PMID 26912385
- [Background] Manzanares J, Julian M, Carrascosa A. Role of the cannabinoid system in pain control and therapeutic implications for the management of acute and chronic pain episodes. Curr Neuropharmacol. 2006 Jul;4(3):239-57. doi: 10.2174/157015906778019527. PMID 18615144
- [Background] Vigil JM, Stith SS, Adams IM, Reeve AP. Associations between medical cannabis and prescription opioid use in chronic pain patients: A preliminary cohort study. PLoS One. 2017 Nov 16;12(11):e0187795. doi: 10.1371/journal.pone.0187795. eCollection 2017. PMID 29145417
- [Background] Lucas P, Walsh Z. Medical cannabis access, use, and substitution for prescription opioids and other substances: A survey of authorized medical cannabis patients. Int J Drug Policy. 2017 Apr;42:30-35. doi: 10.1016/j.drugpo.2017.01.011. Epub 2017 Feb 9. PMID 28189912